CLINICAL TRIAL: NCT03274128
Title: Evaluation of the Effectiveness of Spa Treatment in Swieradow Zdroj With Special Regard to the Action of Radon Waters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wroclaw Medical University (Other)
Responsible Party: Principal Investigator, Jadwiga Kuciel-Lewandowska, Doctor of Medicine, Wroclaw Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KLASTER - 3/2014
Record Dates: First submitted 2017-08-31; First posted 2017-09-06 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Osteoarthritis; Degenerative Disc Disease
MeSH Terms: conditions — Osteoarthritis; Intervertebral Disc Degeneration | interventions — Inhalation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Active Comparator): The treatment included a comprehensive therapy: radon therapeutic baths and inhalations, kinesiotherapy. On the day of admission to the SPA the patients were subjected to subjective and objective examination. Laboratory tests (lipids profile, CRP, smear blood morphology, TAS- total antioxidative potential, metalloproteinase 8) were performed before treatment on day 5 and after 18 days. In addition, before and after treatment, standard scales were used to assess pain intensity: MCGill scale and VAS scale and anxiety and depression levels - HADS scale.
  Interventions: Radiation: Radon therapeutic baths and inhalations; Procedure: Kinesiotherapy
- Control Group (No Intervention): On the day of admission to the SPA the patients were subjected to subjective and objective examination. Laboratory tests (lipids profile, CRP, smear blood morphology, TAS- total antioxidative potential, metalloproteinase 8) were performed before treatment on day 5 and after 18 days. In addition, before and after treatment, standard scales were used to assess pain intensity: MCGill scale and VAS scale and anxiety and depression levels - HADS scale.

INTERVENTIONS:
Radiation: Radon therapeutic baths and inhalations — The natural water with low mineralized content plays a major therapeutic role with the parameters of Rn 303,1-441,5 Bq/l. In the treatment rooms (inhalation, cabins with baths and swimming pool) measurement of alpha radiation was 184,4-450,0 MeV. The measurements were analyzed every 3 months at the Institute of Occupational Medicine in the Department of Radiation Protection in Lodz, Poland. Among the types of treatments used in the therapy there was: comprehensive radon bath - with the temperature of 37 °C, duration 15 min., the treatments were performed every 2nd day, whereas radon inhalations lasted 15 min. with the temp. 37 °C- treatments were performed every 2nd day from Monday to Friday. Baths and inhalations were performed interchangeably and the total number of radon treatments during one stay was 15.
  Arms: Study Group
Procedure: Kinesiotherapy — It is the therapeutic treatment of disease by passive and active muscular movements (as by massage) and of exercise. It is the core element of physiotherapy/physical therapy. Kinesiotherapy - duration of 30-45 min,
  Arms: Study Group

SUMMARY:
Observation conducted during the 21 days of treatment in the health resort of Swieradow-Zdroj. In a treatment of applied therapy: radon therapeutic baths and inhalations, kinesiotherapy. Study group with degenerative joints and disc disease participating in therapy. The control group was selected by the spa workers, also suffering from a degenerative disease of the movement organs not using the spa's treatment base. In both of these groups, appropriate pre- and post-treatment studies were performed.

DETAILED DESCRIPTION:
The observation was conducted during 21 days of medicinal stays in the health resort of Swieradow-Zdroj. The treatment included a comprehensive therapy: radon therapeutic baths and inhalations, kinesiotherapy.

The study group consisted of patients with degenerative joints and disc disease participating in therapy. On the day of admission to the SPA the patients were subjected to subjective and objective examination. Laboratory tests (lipids profile, CRP, smear blood morphology, TAS- total antioxidative potential, metalloproteinase 8) were performed before treatment on day 5 and after 18 days. In addition, before and after treatment, standard scales were used to assess pain intensity: MCGill scale and VAS scale and anxiety and depression levels - HADS scale.

The control group was selected by the spa workers, also suffering from a degenerative disease of the movement organs not using the spa's treatment base. In this group also made the same study.

ELIGIBILITY:
Inclusion Criteria:

* the presence of degenerative joints and/or disc disease;
* age range 40-60 years;
* the written consent to participate in research;
* no impediment to comprehensive treatment at the spa.

Exclusion Criteria:

* the lack of consent to participate in research;
* the age under 40 and over 60 years;
* the presence of diseases constituting a contraindication to therapy (compatible with the standard list of indications and contraindications to spa therapy);
* the presence of metabolic diseases.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2015-04-30 (Actual); Study Completion 2016-03-30 (Actual)

PRIMARY OUTCOMES:
Change of results Laboratory tests (lipids profile, CRP, smear blood morphology, TAS- total antioxidative potential, metalloproteinase 8) on day 5 and after 18 days of therapy | on day 5 and after 18 days of therapy
  The biological material was taken with sterile disposable equipment. After 10 ml of venous blood was collected in a closed system, local laboratory tests were performed, such as morphology with smear, CRP, glycemic control, and lipids profile. Tested using standard tests. Subsequently, 5 ml of venous blood also collected in the closed system directly into the monoveta was centrifuged to obtain serum - a sample to be tested for TAS. Another 5 ml of venous blood collected in the closed system will be left to solidify - sample for metalloproteinase 8. Both specimens were transported at +6 ° C. Analyzes carried out by non-standard and non-commercial laboratory tests serving exclusively for scientific research in the Department of Medical Analyzes of the Medical University of Wroclaw.

SECONDARY OUTCOMES:
Pain Index | on day 5 and after 18 days
  MCGill scale (The McGill Pain Questionnaire) It is a scale of rating pain developed at McGill University by Melzack and Torgerson in 1971. It is a self-report questionnaire that allows individuals to give their doctor a good description of the quality and intensity of pain that they are experiencing. Users first select a single word from each group that best reflects their pain. Users then review the list and select the three words from groups 1-10 that best describe their pain, two words from groups 11-15, a single word from group 16, and then one word from groups 17-20. After completing the questionnaire, users will have selected seven words that best describe their pain. Users can use some words more than once.
Pain Index | on day 5 and after 18 days
  VAS scale (The visual analogue scale) It is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured. When responding to a VAS item, respondents specify their level of agreement to a statement by indicating a position along a continuous line between two end-points. This continuous (or "analogue") aspect of the scale differentiates it from discrete scales such as the Likert scale. There is evidence showing that visual analogue scales have superior metrical characteristics than discrete scales, thus a wider range of statistical methods can be applied to the measurements.
Anxiety and Depression Index | on day 5 and after 18 days
  HADS scale (Hospital Anxiety and Depression Scale) It was originally developed by Zigmond and Snaith (1983)and is commonly used by doctors to determine the levels of anxiety and depression that a patient is experiencing. The HADS is a fourteen item scale that generates ordinal data. Seven of the items relate to anxiety and seven relate to depression. Zigmond and Snaith created this outcome measure specifically to avoid reliance on aspects of these conditions that are also common somatic symptoms of illness, for example fatigue and insomnia or hypersomnia. This, it was hoped, would create a tool for the detection of anxiety and depression in people with physical health problems.

CONTACTS AND LOCATIONS:
Overall Officials: Jadwiga Kuciel-Lewandowska, MD, Study Director — MD, Departament of Spa Treatment, History Physical Medicine and Balneology Medical University of Wroclaw

IPD SHARING:
Plan to Share IPD: Undecided
Any request to share the IPD will be considered individually and in the group of all researchers who have participated in the research. Due to the law at the Medical University of Wroclaw every interested IPD of our study must also write a request to the Deputy Dean for the University of Medicine in Wroclaw to obtain access to such documents from him. The applicant will receive all contact details for the Deputy Dean for the University of Medical in Wroclaw when applying for access to the IPD.

REFERENCES:
- [Derived] Kuciel-Lewandowska J, Kasperczak M, Pawlik-Sobecka L, Paprocka-Borowicz M, Gnus J. Assessment of Changes in Concentration of Total Antioxidant Status, Acute-Phase Protein, and Prolactin in Patients with Osteoarthritis Subjected to a Complex Spa Treatment with Radon Water: Preliminary Results. PPAR Res. 2020 Apr 23;2020:9459418. doi: 10.1155/2020/9459418. eCollection 2020. PMID 32373171
- [Derived] Kasperczak M, Kuciel-Lewandowska J, Gnus J, Paprocka-Borowicz M. Assessment of Changes in Lipids Metabolism in Patients with Degenerative Joints and Discs Diseases Subjected to Spa Therapy. Biomed Res Int. 2019 Jul 24;2019:4732654. doi: 10.1155/2019/4732654. eCollection 2019. PMID 31428637
- [Derived] Kuciel-Lewandowska J, Gnus J, Pawlik-Sobecka L, Placzkowska S, Kokot I, Kasperczak M, Paprocka-Borowicz M. The Assessment of the Integrated Antioxidant System of the Body in the Course of Radon Therapy: A Pilot Study. Biomed Res Int. 2018 Jan 2;2018:6038106. doi: 10.1155/2018/6038106. eCollection 2018. PMID 29487870